CLINICAL TRIAL: NCT05200455
Title: Microelectrodes in Epilepsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Barbara Jobst, Chair, Department of Neurology, Dartmouth-Hitchcock Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STUDY00021993; 1R01NS074450-01 (NIH)
Record Dates: First submitted 2022-01-07; First posted 2022-01-20 (Actual); Results first posted 2022-09-07 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-08

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy | interventions — Microelectrodes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Microelectrodes (Experimental): Patients who qualify for this study will be implanted with standard electrodes as well as microelectrodes for their intracranial seizure monitoring.
  Interventions: Device: Microelectrodes

INTERVENTIONS:
Device: Microelectrodes — Microelectrode implantation

SUMMARY:
The purpose of this study is to test microelectrodes in intracranial monitoring to see if they will provide novel information on the epileptic potential of the implanted brain tissue. A secondary objective is to investigate the activity of single neurons during specific cognitive tasks.

DETAILED DESCRIPTION:
The standard-of-care for medically refractory epilepsy is resective brain surgery. In certain patients, precise localization of the epileptic focus is done using intracranial EEG (iEEG) recording. In this type of EEG recording, electrodes are placed on the brain surface or inserted into the brain through an opening in the skull. In addition to standard electrode recording, this study will use ultra thin microelectrodes. Microelectrodes are only several micrometers thick and are useful because they are able to record the activity of single neurons in isolation. Such recordings have tremendous clinical potential in epilepsy surgery and tremendous research potential in cognitive neuroscience.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 year old
* male or female
* right or left handed
* IQ>70
* medically refractory focal epilepsy requiring intracranial EEG for pre-surgical evaluation deemed medically necessary
* no contraindications to intracranial electrode study
* able and willing to participate in research

Exclusion Criteria:

* does not meet the inclusion criteria

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2009-09-18 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-05-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara C Jobst, MD, PhD, Principal Investigator — Section Chief of Adult Neurology
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Microelectrodes: Patients who qualify for this study were implanted with standard electrodes that in addition have microelectrodes embedded in the standard macroelectrodes that are standard of care in epilepsy surgery. Microelectrodes have been shown to record single unit potentials and more localized field potentials on EEG recordings. There is no control group as patient serve as their own control. The patient is presented with a cognitive task and signals are recorded during the cognitive task, the signals during the different elements of the cognitive task are compared to each other or compared to a baseline state.
  There is no therapeutic intervention tested, the study is aimed to understand cognitive memory processing and translate animal studies to humans that have described successful memory encoding with certain EEG signals (place cells, theta oscillations)
Period: Overall Study
Arm/Group | Microelectrodes
Started | 34
Completed | 30
Not Completed | 4
Not completed — These patients were not implanted with intracranial electrodes for clinical reasons . | 4

BASELINE CHARACTERISTICS:
Arm/Group | Microelectrodes
Number analyzed (Participants) | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 34
  >=65 years | 0
Sex/Gender, Customized [Count of Participants; unit: Participants] | 34
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 33
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Microelectrode Technology to Isolate Place Responsive Neurons in the Human Hippocampus as Measured by the Number of Place Responsive Neurons.
Description: With the occipito-temporal implantation approach of implantation of microelectrodes, feasibility will measured by the number of place responsive neurons that could be isolated.
Time Frame: Evaluated for each patient during monitoring period of approximately 2 weeks
Population: Participants included patients undergoing intra-cranial EEG monitoring for TLE and are implanted with depth electrodes and microelectrodes via the trans-occipital approach. The total number of place responsive neurons recorded from all participants is reported below.
Measure: Number; unit: place responsive neurons
Arm/Group | Microelectrodes
Number analyzed (Participants) | 30
place responsive neurons | 79

2. Secondary Outcome: How Precise the Frequencies (Alpha, Beta, Delta, Theta, Gamma, and High-gamma) of Neural Brain Activity Predict the Speed of the Participant at Performing the Cognitive Task (Accuracy Measured in Percentage).
Description: Secondary objective is to investigate whether it is possible to predict the speed of which each participant is performing and navigating during the cognitive task via the intracranial spectral EEG changes (alpha, beta, delta, theta, gamma, and high-gamma) during these tasks. Accuracy of frequency band (brain waves) predicting speed during specific cognitive tasks is measured by how precisely the frequency band predicts navigational speed and is expressed as a percentage of correct prediction.
Time Frame: Evaluated for each patient during monitoring period of approximately 2 weeks
Population: Participants included patients undergoing intra-cranial EEG monitoring for TLE and are implanted with depth electrodes and microelectrodes.
Measure: Mean (Inter-Quartile Range); unit: percentage of accuracy in decimals
Groups:
- Microelectrodes: Participants included patients undergoing intra-cranial EEG monitoring for temporal lobe epilepsy and are implanted with depth electrodes and microelectrodes.
Arm/Group | Microelectrodes
Number analyzed (Participants) | 30
percentage of accuracy in decimals
  Delta | 0.477 [0.400 to 0.492]
  Theta | 0.490 [0.449 to 0.499]
  Alpha | 0.440 [0.372 to 0.477]
  Beta | 0.444 [0.388 to 0.537]
  Gamma | 0.362 [0.290 to 0.419]
  High-gamma | 0.382 [0.305 to 0.405]

ADVERSE EVENTS:
Time Frame: Evaluated for each patient during monitoring period of approximately 2 weeks
Arm/Group | Microelectrodes
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 2/30
Other Adverse Events (participants affected / at risk) | 0/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Microelectrodes (N=30)
Infection (Infections and infestations) | 1 (1) — Subject had post operative wound infection following craniotomy. This was recorded as a serious adverse event that was unrelated to the study procedure.
Chronic Inflammatory Reaction (Infections and infestations) | 1 (1) — Study subject had fever of unknown etiology, cerebritis, chronic inflammatory reaction. This was recorded as a serious adverse event that was unrelated to the study procedure.

LIMITATIONS AND CAVEATS:
Too few single units were recorded, and it was not possible to identify the units as place cells.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-06-22): https://cdn.clinicaltrials.gov/large-docs/55/NCT05200455/Prot_SAP_000.pdf
  • Informed Consent Form (2014-06-19): https://cdn.clinicaltrials.gov/large-docs/55/NCT05200455/ICF_001.pdf